CLINICAL TRIAL: NCT02047708
Title: A Phase II, Single Centre, Randomised, Placebo-controlled, 3-part Trial to Assess the Safety, Tolerability and Efficacy of Zibotentan in Patients With Renal Disease Secondary to Scleroderma
Brief Title: Zibotentan Better Renal Scleroderma Outcome Study
Acronym: ZEBRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-003200-39
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Scleroderma; Scleroderma Renal Crisis; Chronic Kidney Disease
MeSH Terms: conditions — Scleroderma, Diffuse; Renal Insufficiency, Chronic | interventions — ZD4054

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Zibotentan — Selective endothelin-A antagonist
  Other Names: ZD4054

SUMMARY:
Many patients with scleroderma have damage to their kidneys caused by the disease. There is limited evidence for treatments to prevent this damage or stop it progressing. Blocking a substance in the blood called endothelin has helped treat some aspects of scleroderma. The purpose of this study is to see how effective a new endothelin blocker called Zibotentan is in treating patients who have scleroderma and have gone on to develop reduced kidney function as a complication. It will be given in addition to the accepted treatments used for scleroderma. There will be three parts to this study each for a different group of patients:

* ZEBRA 1 for patients with mild or moderate kidney disease caused by scleroderma
* ZEBRA 2A for patients with a more severe, acute form of kidney disease caused by scleroderma (scleroderma renal crisis) who do not require dialysis
* ZEBRA 2B for patients who have had scleroderma renal crisis and are on dialysis

DETAILED DESCRIPTION:
This is a 3-part study (Zebra 1, 2A and 2B) that will explore safety and therapeutic potential of Zibotentan in acute and chronic renal complications of Scleroderma. Trial duration will be 52 weeks for Zebra 1 and 2A (1 or 2 weeks for ZEBRA 2B with 1 year follow up data). Scleroderma (Systemic sclerosis) is a multisystem rheumatic disease that results in vascular damage and fibrosis of target organs.This project will focus specifically on the evaluation and treatment of renal disease in scleroderma.

Renal involvement in Scleroderma occurs with a variety of different pathologies; hypertensive scleroderma renal crisis (SRC) being the most dramatic manifestation but milder forms of chronic renal disease are frequent and represent an important clinical feature.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with scleroderma and:
2. CKD 2/3 (ZEBRA 1)
3. Renal crisis not on dialysis (ZEBRA 2A)
4. Renal crisis on dialysis (ZEBRA 2B)

Exclusion Criteria:

1. Previous use of an endothelin receptor antagonist within 3 months of the study start
2. Significant abnormalities in liver function testing (ALT, ALP, Bilirubin) more than three times upper limit of normal)
3. Patients with body weight <40kg.
4. Patients with conditions which prevent compliance with the protocol or failure to adhere to therapy.
5. Patients with any other life threatening condition.
6. Patients with known hypersensitivity to Zibotentan or its excipients
7. Previous history of epilepsy or other CNS AEs, neurologic symptoms or signs consistent with acute or evolving spinal cord compression, and CNS metastases
8. Patients with a baseline left ventricular ejection fraction < 40% (prior to any scleroderma renal crisis), patients with acute myocardial infarction within six months or patients who are judged by the trial clinician to be at unacceptable risk from cardiac complications.
9. History of chronic alcohol or drug abuse or any condition associated with poor compliance as judged by the investigator
10. Patients receiving cyclosporin A within 1 week of screening or expecting to receive this agent during the study.
11. Patients who have received an investigational agent in the month prior to screening. These patients may be eligible if after a month of washout period, they are still within 112 months of the onset of the Scleroderma renal crisis.
12. Active malignancy or neoplastic disease in the previous 12 months
13. Women who rely on oestrogencontaining contraceptives (due to potential drug interaction with Zibotentan).
14. Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
sVCAM 1 soluble Vascular Cell Adhesion Molecule | 12 months
  sVCAM1 is a biomarker of renal involvement in scleroderma

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Stern EP, Host LV, Wanjiku I, Escott KJ, Gilmour PS, Ochiel R, Unwin R, Burns A, Ong VH, Cadiou H, O'Keeffe AG, Denton CP. Zibotentan in systemic sclerosis-associated chronic kidney disease: a phase II randomised placebo-controlled trial. Arthritis Res Ther. 2022 Jun 1;24(1):130. doi: 10.1186/s13075-022-02818-6. PMID 35650639